CLINICAL TRIAL: NCT06796972
Title: In Utero Surgery for Fetal Myelomeningocele: Decision-making Mechanisms and Psychological Impact of Prenatal Therapy
Acronym: PriumPsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP230369
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Myelomeningocele
Keywords: Psychology; fetal myelomeningocele; Parents
MeSH Terms: conditions — Meningomyelocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Parents of children operated on in utero (Other): Semi-structured interviews with a psychologist
  Interventions: Other: Semi-structured interviews with a psychologist

INTERVENTIONS:
Other: Semi-structured interviews with a psychologist — Semi-directed interviews using an interview guide on different themes

SUMMARY:
Myelomeningocele is a malformation of the spine and spinal cord, generally diagnosed prenatally, and responsible for a complex disability for the unborn child. In the event of continued pregnancy, in utero surgery can be performed to improve the prognosis of the children. This fetal therapy does not allow a cure and induces risks for the fetus, and for the mother, both during surgery and for her obstetric future.

Currently, few studies have focused on the factors influencing the choice to resort to in utero surgery and the experience of patients and co-parents before and after this intervention. No qualitative study on the subject has been published to date.

DETAILED DESCRIPTION:
The study population corresponds to all couples who have chosen to continue the pregnancy in the face of a prenatal diagnosis of myelomeningocele in their fetus as well as to resort to in utero surgery to repair this malformation. In order to obtain the largest possible sample, the study will be offered to both couples who have had open surgery and those who have had fetoscopy.

This study aims to investigate, a posteriori, the experience of couples who have chosen fetal surgery to repair a myelomeningocele.

This is a study in clinical psychology, cross-sectional observational with an approach that will be mixed, qualitative and quantitative.

In practice, the only procedures added by the research will consist of:

* an interview between the mother of the child operated on in utero and a psychologist researcher-student pair in Master 2 of psychology
* an interview between the father of the child operated on in utero and a psychologist researcher-student pair in Master 2 of psychology
* the completion of a decision scale by each of the parents The presence of the interview with a psychologist not planned as part of the care may lead to the modification of the usual care of the parents.

ELIGIBILITY:
Inclusion Criteria:

* Mothers and adult co-parents of the child with MMC operated in utero, having signed informed consent. If both members of the couple have agreed to participate, they will be received separately.
* Mother who had fetal surgery for in utero repair of a fetal myelomeningocele by laparotomy and hysterotomy aged 18 years or older at the time of surgery, and whose child affected by the surgery is at least 6 months old
* Speaking French
* Not presenting a severe psychiatric disorder altering the relationship with reality
* Patient affiliated to a social security system

Exclusion Criteria:

* Patient under guardianship or curatorship, deprived of liberty or unable to sign informed consent to participate in the study
* Patient under State Medical Aid

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Studying the experience of couples who have chosen fetal surgery | up to 18 months
  Semi-structured interviews with a psychologist

SECONDARY OUTCOMES:
Investigate the decision-making factors that contributed to the choice of prenatal surgery | Up to 18 months
  Semi-structured interviews with a psychologist
Evaluate the quality of the information that couples received regarding the three possibilities proposed when faced with a prenatal diagnosis of myelomeningocele | Up to 18 months
  Semi-structured interviews with a psychologist

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine Foetale Hôpital Armand Trousseau, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No